CLINICAL TRIAL: NCT02854527
Title: Investigation of Mutual Pharmacokinetic Interactions of Digoxin, Furosemide, Metformin, and Rosuvastatin Given All Together as a Probe Cocktail for Key Drug Transporters (an Open-label, Randomised, Single-dose, Five-way Crossover Study)
Brief Title: Transporter Cocktail Mutual Interaction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 352.2096; 2016-001893-14 (EudraCT Number)
Record Dates: First submitted 2016-08-01; First posted 2016-08-03 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — Digoxin; Furosemide; Metformin; Rosuvastatin Calcium

ARMS (5):
- R1 (Reference 1) Digoxin (Experimental): 1 tablet (0.25 mg) digoxin as single dose
  Interventions: Drug: Digoxin
- R2 Furosemide (Experimental): 0.1 mL (1 mg) furosemide oral solution as single dose
  Interventions: Drug: Furosemide
- R3 Metformin hydrochloride (Experimental): 0.1 mL (10 mg) metformin oral solution as single dose
  Interventions: Drug: Metformin
- R4 Rosuvastatin (Experimental): 1 tablet (10 mg) rosuvastatin as single dose
  Interventions: Drug: Rosuvastatin
- T (Test) (Experimental): 1 tablet (0.25 mg) digoxin, 0.1 mL (1 mg) furosemide oral solution, 0.1 mL (10 mg) metformin oral solution, and 1 tablet (10 mg) rosuvastatin, all together as a single dose ('cocktail')
  Interventions: Drug: Digoxin; Drug: Furosemide; Drug: Metformin hydrochloride; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Digoxin — single dose
  Arms: R1 (Reference 1) Digoxin
Drug: Furosemide — single dose
  Arms: R2 Furosemide
Drug: Metformin — single dose
  Arms: R3 Metformin hydrochloride
Drug: Rosuvastatin — single dose
  Arms: R4 Rosuvastatin
Drug: Digoxin — 0.25 mg digoxin as single dose (all 4 drugs given together as a cocktail at the same time point)
  Arms: T (Test)
Drug: Furosemide — 1 mg furosemide as single dose (all 4 drugs given together as a cocktail at the same time point)
  Arms: T (Test)
Drug: Metformin hydrochloride — 10 mg metformin hydrochloride as single dose (all 4 drugs given together as a cocktail at the same time point)
  Arms: T (Test)
Drug: Rosuvastatin — 10 mg rosuvastatin as single dose (all 4 drugs given together as a cocktail at the same time point)
  Arms: T (Test)

SUMMARY:
Main objective is to investigate mutual pharmacokinetic drug-drug interactions of digoxin, furosemide, metformin, and rosuvastatin when given all together as a cocktail

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and local legislation

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients, sulphonamides, or cardiac glycosides)
* Use of drugs within 30 days prior to administration of trial medication that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation (corrected Q-T interval)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

* Hypokalemia, hypomagnesemia, or hypercalcemia
* PQ ( (time between the onset of the P wave (atrial activity) and the QRS complex (ventricular activity)) interval greater than 220 ms in the ECG at screening
* Myopathy
* Hereditary galactose or fructose intolerance, lactase deficiency, or glucose-galactose malabsorption

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is an open-label, randomised, single-dose, five-way, ten-sequence crossover study. Four drugs (Digoxin (R1), Furosemide, (R2), Metformin hydrochloride (R3), Rosuvastatin (R4)) were given as monotherapy and one as a combination of all four drugs together as test cocktail (T) in pre-defined sequences.
Groups:
- ABECD (R1->R2->T->R3->R4): Subjects in this sequence were administered five different treatments in a sequence with a washout period of at least 10 days between each drug administration of adjacent treatment periods. First, they were administered a single dose of 0.25 milligram (mg) tablet of Digoxin (reference 1 or R1). Second, they were administered a single dose of 0.1 milliliter (mL) or 1 mg oral solution of Furosemide (R2). Third, they were administered a single dose of test cocktail (T) comprised of 0.25 mg of Digoxin, 0.1 mL (1 mg) of Furosemide, 0.1 mL (10 mg) of Metformin hydrochloride and 10 mg of Rosuvastatin. Fourth, they were administered a single dose of 0.1 mL (10 mg) oral solution of Metformin hydrochloride (R3). Fifth, they were administered a single dose of 10 mg film-coated tablet of Rosuvastatin (R4).
  All drugs were administered orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
- AEBDC (R1->T->R2->R4->R3): Subjects in this sequence were administered five different treatments in a sequence with a washout period of at least 10 days between each drug administration of adjacent treatment periods. First, they were administered a single dose of 0.25 milligram (mg) tablet of Digoxin (reference 1 or R1). Second, they were administered a single dose of test cocktail (T) comprised of 0.25 mg of Digoxin, 0.1 mL (1 mg) of Furosemide, 0.1 mL (10 mg) of Metformin hydrochloride and 10 mg of Rosuvastatin. Third, they were administered a single dose of 0.1 milliliter (mL) or 1 mg oral solution of Furosemide (R2). Fourth, they were administered a single dose of 10 mg film-coated tablet of Rosuvastatin (R4). Fifth, they were administered a single dose of 0.1 mL (10 mg) oral solution of Metformin hydrochloride (R3).
  All drugs were administered orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
- BACED (R2->R1->R3->T->R4): Subjects in this sequence were administered five different treatments in a sequence with a washout period of at least 10 days between each drug administration of adjacent treatment periods. First, they were administered a single dose of 0.1 milliliter (mL) or 1 mg oral solution of Furosemide (reference 2 or R2). Second, they were administered a single dose of 0.25 milligram (mg) tablet of Digoxin (R1). Third, they were administered a single dose of 0.1 mL (10 mg) oral solution of Metformin hydrochloride (R3). Fourth, they were administered a single dose of test cocktail (T) comprised of 0.25 mg of Digoxin, 0.1 mL (1 mg) of Furosemide, 0.1 mL (10 mg) of Metformin hydrochloride and 10 mg of Rosuvastatin. Fifth, they were administered a single dose of 10 mg film-coated tablet of Rosuvastatin (R4).
  All drugs were administered orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
- BCADE (R2->R3->R1->R4->T): Subjects in this sequence were administered five different treatments in a sequence with a washout period of at least 10 days between each drug administration of adjacent treatment periods. First, they were administered a single dose of 0.1 milliliter (mL) or 1 mg oral solution of Furosemide (R2). Second, they were administered a single dose of 0.1 mL (10 mg) oral solution of Metformin hydrochloride (R3). Third, they were administered a single dose of 0.25 milligram (mg) tablet of Digoxin (R1). Fourth, they were administered a single dose of 10 mg film-coated tablet of Rosuvastatin (R4). Fifth, they were administered a single dose of test cocktail (T) comprised of 0.25 mg of Digoxin, 0.1 mL (1 mg) of Furosemide, 0.1 mL (10 mg) of Metformin hydrochloride and 10 mg of Rosuvastatin.
  All drugs were administered orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
- CBDAE (R3->R2->R4->R1->T): Subjects in this sequence were administered five different treatments in a sequence with a washout period of at least 10 days between each drug administration of adjacent treatment periods. First, they were administered a single dose of 0.1 mL (10 mg) oral solution of Metformin hydrochloride (R3). Second, they were administered a single dose of 0.1 milliliter (mL) or 1 mg oral solution of Furosemide (R2). Third, they were administered a single dose of 10 mg film-coated tablet of Rosuvastatin (R4). Fourth, they were administered a single dose of 0.25 milligram (mg) tablet of Digoxin (R1). Fifth, they were administered a single dose of test cocktail (T) comprised of 0.25 mg of Digoxin, 0.1 mL (1 mg) of Furosemide, 0.1 mL (10 mg) of Metformin hydrochloride and 10 mg of Rosuvastatin.
  All drugs were administered orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
- CDBEA (R3->R4->R2->T->R1): Subjects in this sequence were administered five different treatments in a sequence with a washout period of at least 10 days between each drug administration of adjacent treatment periods. First, they were administered a single dose of 0.1 mL (10 mg) oral solution of Metformin hydrochloride (R3). Second, they were administered a single dose of 10 mg film-coated tablet of Rosuvastatin (R4). Third, they were administered a single dose of 0.1 milliliter (mL) or 1 mg oral solution of Furosemide (R2). Fourth, they were administered a single dose of test cocktail (T) comprised of 0.25 mg of Digoxin, 0.1 mL (1 mg) of Furosemide, 0.1 mL (10 mg) of Metformin hydrochloride and 10 mg of Rosuvastatin. Fifth, they were administered a single dose of 0.25 milligram (mg) tablet of Digoxin (R1).
  All drugs were administered orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
- DCEBA (R4->R3->T->R2->R1): Subjects in this sequence were administered five different treatments in a sequence with a washout period of at least 10 days between each drug administration of adjacent treatment periods. First, they were administered a single dose of 10 mg film-coated tablet of Rosuvastatin (R4). Second, they were administered a single dose of 0.1 mL (10 mg) oral solution of Metformin hydrochloride (R3). Third, they were administered a single dose of test cocktail (T) comprised of 0.25 mg of Digoxin, 0.1 mL (1 mg) of Furosemide, 0.1 mL (10 mg) of Metformin hydrochloride and 10 mg of Rosuvastatin. Fourth, they were administered a single dose of 0.1 milliliter (mL) or 1 mg oral solution of Furosemide (R2). Fifth, they were administered a single dose of 0.25 milligram (mg) tablet of Digoxin (R1).
  All drugs were administered orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
- DECAB (R4->T->R3->R1->R2): Subjects in this sequence were administered five different treatments in a sequence with a washout period of at least 10 days between each drug administration of adjacent treatment periods. First, they were administered a single dose of 10 mg film-coated tablet of Rosuvastatin (R4). Second, they were administered a single dose of test cocktail (T) comprised of 0.25 mg of Digoxin, 0.1 mL (1 mg) of Furosemide, 0.1 mL (10 mg) of Metformin hydrochloride and 10 mg of Rosuvastatin. Third, they were administered a single dose of 0.1 mL (10 mg) oral solution of Metformin hydrochloride (R3). Fourth, they were administered a single dose of 0.25 milligram (mg) tablet of Digoxin (R1). Fifth, they were administered a single dose of 0.1 milliliter (mL) or 1 mg oral solution of Furosemide (R2).
  All drugs were administered orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
- EADBC (T->R1->R4->R2->R3): Subjects in this sequence were administered five different treatments in a sequence with a washout period of at least 10 days between each drug administration of adjacent treatment periods. First, they were administered a single dose of test cocktail (T) comprised of 0.25 mg of Digoxin, 0.1 mL (1 mg) of Furosemide, 0.1 mL (10 mg) of Metformin hydrochloride and 10 mg of Rosuvastatin. Second, they were administered a single dose of 0.25 milligram (mg) tablet of Digoxin (R1). Third, they were administered a single dose of 10 mg film-coated tablet of Rosuvastatin (R4). Fourth, they were administered a single dose of 0.1 milliliter (mL) or 1 mg oral solution of Furosemide (R2). Fifth, they were administered a single dose of 0.1 mL (10 mg) oral solution of Metformin hydrochloride (R3).
  All drugs were administered orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
- EDACB (T->R4->R1->R3->R2): Subjects in this sequence were administered five different treatments in a sequence with a washout period of at least 10 days between each drug administration of adjacent treatment periods. First, they were administered a single dose of test cocktail (T) comprised of 0.25 mg of Digoxin, 0.1 mL (1 mg) of Furosemide, 0.1 mL (10 mg) of Metformin hydrochloride and 10 mg of Rosuvastatin. Second, they were administered a single dose of 10 mg film-coated tablet of Rosuvastatin (R4). Third, they were administered a single dose of 0.25 milligram (mg) tablet of Digoxin (R1). Fourth, they were administered a single dose of 0.1 mL (10 mg) oral solution of Metformin hydrochloride (R3). Fifth, they were administered a single dose of 0.1 milliliter (mL) or 1 mg oral solution of Furosemide (R2).
  All drugs were administered orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
Period: Overall Study
Arm/Group | ABECD (R1->R2->T->R3->R4) | AEBDC (R1->T->R2->R4->R3) | BACED (R2->R1->R3->T->R4) | BCADE (R2->R3->R1->R4->T) | CBDAE (R3->R2->R4->R1->T) | CDBEA (R3->R4->R2->T->R1) | DCEBA (R4->R3->T->R2->R1) | DECAB (R4->T->R3->R1->R2) | EADBC (T->R1->R4->R2->R3) | EDACB (T->R4->R1->R3->R2)
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Received R1 | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Received R2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Received R3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3
Received R4 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3
Received T | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The randomised set (RS) included all randomised subjects, whether treated or not
Groups:
- Total: Total of all reporting groups
Arm/Group | ABECD (R1->R2->T->R3->R4) | AEBDC (R1->T->R2->R4->R3) | BACED (R2->R1->R3->T->R4) | BCADE (R2->R3->R1->R4->T) | CBDAE (R3->R2->R4->R1->T) | CDBEA (R3->R4->R2->T->R1) | DCEBA (R4->R3->T->R2->R1) | DECAB (R4->T->R3->R1->R2) | EADBC (T->R1->R4->R2->R3) | EDACB (T->R4->R1->R3->R2) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.7 (2.5) | 28.7 (8.1) | 41.3 (15.8) | 42.0 (5.3) | 32.3 (9.0) | 45.7 (7.2) | 30.3 (6.4) | 33.0 (9.6) | 40.3 (7.5) | 34.3 (7.2) | 35.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 30

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of Digoxin From 0 to Last Quantifiable Data Point (AUC 0-tz)
Description: Area under the concentration-time curve of digoxin in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz). Standard error presented is actually geometric standard error. CI - confidence interval, gMean - geometric mean.
Time Frame: Blood sampling at 2:00 (hour: minute) before drug administration, 0:20, 0:40, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 10:00, 12:00, 24:00, 36:00, 48:00, 72:00 and 96:00 after drug administration
Population: The Pharmacokinetic (PK) analysis set (PKS) included all randomized subjects who were documented to have taken at least 1 dose of study drug and who have provided at least 1 primary or secondary PK endpoint that was not excluded from analysis due to non-evaluability or protocol violation relevant for the evaluation of the pharmacokinetics.
Measure: Geometric Mean (Standard Error); unit: nanomole hour per liter (nmol·h/L)
Groups:
- Test Cocktail (T): Subjects were administered a single dose of test cocktail (T) comprised of 0.25 mg tablet of Digoxin, 0.1 mL (1 mg) oral solution of Furosemide, 0.1 mL (10 mg) oral solution of Metformin hydrochloride and 10 mg film-coated tablet of Rosuvastatin orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
- Digoxin (R1): Subjects were administered a single dose of 0.25 milligram (mg) tablet of Digoxin orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
Arm/Group | Test Cocktail (T) | Digoxin (R1)
Number analyzed (Participants) | 28 | 28
nanomole hour per liter (nmol·h/L) | 11.549 (1.053) | 11.981 (1.053)
Statistical Analysis 1: Comparison: Test Cocktail (T) vs Digoxin (R1); This statistical analysis assess the effect of the other cocktail compounds in treatment T on the first primary outcome measure of treatment R1; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects: 'sequence', 'subject within sequence', 'period' and 'treatment'; Adjusted Geometric mean ratio (T/R1) (%) = 96.39, 90% CI 2-sided [88.22 to 105.33], Standard Deviation 19.4 — Least square estimates of log-transformed PK endpoint for T and R1 were back transformed to original scale to get adjusted gMean ratio (T/R1) and its 2-sided 90% CI. Standard deviation is intra-individual geometric coefficient of variation (%)

2. Primary Outcome: Maximum Concentration of Digoxin (Cmax)
Description: This outcome measure presents the maximum measured concentration of digoxin in plasma (Cmax). Standard error presented is actually geometric standard error.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nanomole per liter (nmol/L)
Arm/Group | Test Cocktail (T) | Digoxin (R1)
Number analyzed (Participants) | 28 | 28
nanomole per liter (nmol/L) | 1.262 (1.047) | 1.355 (1.047)
Statistical Analysis 1: Comparison: Test Cocktail (T) vs Digoxin (R1); This statistical analysis assess the effect of the other cocktail compounds in treatment T on the second primary outcome measure of treatment R1; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric mean ratio (T/R1) (%) = 93.17, 90% CI 2-sided [83.49 to 103.97], Standard Deviation 24.1 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Area Under the Curve of Furosemide From 0 to Last Quantifiable Data Point (AUC 0-tz)
Description: Area under the concentration-time curve of furosemide in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz). Standard error presented is actually geometric standard error.
Time Frame: Blood sampling at 2:00 (hour: minute) before drug administration, 0:20, 0:40, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 10:00, 12:00 and 24:00 after drug administration
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol·h/L
Groups:
- Furosemide (R2): Subjects were administered a single dose of 0.1 milliliter (mL) or 1 mg oral solution of Furosemide orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
Arm/Group | Test Cocktail (T) | Furosemide (R2)
Number analyzed (Participants) | 28 | 30
nmol·h/L | 163.614 (1.039) | 159.434 (1.038)
Statistical Analysis 1: Comparison: Test Cocktail (T) vs Furosemide (R2); This statistical analysis assess the effect of the other cocktail compounds in treatment T on the first primary outcome measure of treatment R2; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric mean ratio (T/R2) (%) = 102.62, 90% CI 2-sided [93.82 to 112.25], Standard Deviation 20.4 — Least square estimates of log-transformed PK endpoint for T and R2 were back transformed to original scale to get adjusted gMean ratio (T/R2) and its 2-sided 90% CI. Standard deviation is intra-individual geometric coefficient of variation (%)

4. Primary Outcome: Maximum Concentration of Furosemide (Cmax)
Description: This outcome measure presents the maximum measured concentration of furosemide in plasma (Cmax). Standard error presented is actually geometric standard error.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol/L
Arm/Group | Test Cocktail (T) | Furosemide (R2)
Number analyzed (Participants) | 28 | 30
nmol/L | 86.275 (1.046) | 82.990 (1.044)
Statistical Analysis 1: Comparison: Test Cocktail (T) vs Furosemide (R2); This statistical analysis assess the effect of the other cocktail compounds in treatment T on the second primary outcome measure of treatment R2; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric mean ratio (T/R2) (%) = 103.96, 90% CI 2-sided [93.60 to 115.46], Standard Deviation 24.0 — [estimate comment as in outcome 3, analysis 1]

5. Primary Outcome: Area Under the Curve of Metformin From 0 to Last Quantifiable Data Point (AUC 0-tz)
Description: Area under the concentration-time curve of metformin in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz). Standard error presented is actually geometric standard error.
Time Frame: Blood sampling at 2:00 (hour: minute) before drug administration, 0:20, 0:40, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 10:00, 12:00, 24:00, 36:00 and 48:00 after drug administration
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol·h/L
Groups:
- Metformin Hydrochloride (R3): Subjects were administered a single dose of 0.1 mL (10 mg) oral solution of Metformin hydrochloride orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
Arm/Group | Test Cocktail (T) | Metformin Hydrochloride (R3)
Number analyzed (Participants) | 28 | 29
nmol·h/L | 1283.797 (1.034) | 1316.790 (1.033)
Statistical Analysis 1: Comparison: Test Cocktail (T) vs Metformin Hydrochloride (R3); This statistical analysis assess the effect of the other cocktail compounds in treatment T on the first primary outcome measure of treatment R3; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric mean ratio (T/R3) (%) = 97.49, 90% CI 2-sided [93.54 to 101.61], Standard Deviation 9.0 — Least square estimates of log-transformed PK endpoint for T and R3 were back transformed to original scale to get adjusted gMean ratio (T/R3) and its 2-sided 90% CI. Standard deviation is intra-individual geometric coefficient of variation (%)

6. Primary Outcome: Maximum Concentration of Metformin (Cmax)
Description: This outcome measure presents the maximum measured concentration of metformin in plasma (Cmax). Standard error presented is actually geometric standard error.
Time Frame: as for outcome 5
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol/L
Arm/Group | Test Cocktail (T) | Metformin Hydrochloride (R3)
Number analyzed (Participants) | 28 | 29
nmol/L | 225.156 (1.045) | 229.171 (1.044)
Statistical Analysis 1: Comparison: Test Cocktail (T) vs Metformin Hydrochloride (R3); This statistical analysis assess the effect of the other cocktail compounds in treatment T on the second primary outcome measure of treatment R3; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric mean ratio (T/R3) (%) = 98.25, 90% CI 2-sided [91.85 to 105.09], Standard Deviation 14.7 — [estimate comment as in outcome 5, analysis 1]

7. Primary Outcome: Area Under the Curve of Rosuvastatin From 0 to Last Quantifiable Data Point (AUC 0-tz)
Description: Area under the concentration-time curve of rosuvastatin in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz). Standard error presented is actually geometric standard error.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol·h/L
Groups:
- Rosuvastatin (R4): Subjects were administered a single dose of 10 mg film-coated tablet of Rosuvastatin orally with 320 mL of non-sparkling drinking water after overnight fasting of 10 hours.
Arm/Group | Test Cocktail (T) | Rosuvastatin (R4)
Number analyzed (Participants) | 28 | 29
nmol·h/L | 81.925 (1.070) | 78.016 (1.069)
Statistical Analysis 1: Comparison: Test Cocktail (T) vs Rosuvastatin (R4); This statistical analysis assess the effect of the other cocktail compounds in treatment T on the first primary outcome measure of treatment R4; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric mean ratio (T/R4) (%) = 105.01, 90% CI 2-sided [96.39 to 114.40], Standard Deviation 18.8 — Least square estimates of log-transformed PK endpoint for T and R4 were back transformed to original scale to get adjusted gMean ratio (T/R4) and its 2-sided 90% CI. Standard deviation is intra-individual geometric coefficient of variation (%)

8. Primary Outcome: Maximum Concentration of Rosuvastatin (Cmax)
Description: This outcome measure presents the maximum measured concentration of rosuvastatin in plasma (Cmax). Standard error presented is actually geometric standard error.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol/L
Arm/Group | Test Cocktail (T) | Rosuvastatin (R4)
Number analyzed (Participants) | 28 | 29
nmol/L | 8.135 (1.074) | 7.801 (1.073)
Statistical Analysis 1: Comparison: Test Cocktail (T) vs Rosuvastatin (R4); This statistical analysis assess the effect of the other cocktail compounds in treatment T on the second primary outcome measure of treatment R4; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric mean ratio (T/R4) (%) = 104.28, 90% CI 2-sided [94.95 to 114.53], Standard Deviation 20.6 — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Area Under the Curve of Digoxin From 0 Extrapolated to Infinity (AUC 0-∞)
Description: Area under the concentration-time curve of digoxin in plasma over the time interval from 0 extrapolated to infinity (AUC 0-∞). Standard error presented is actually geometric standard error.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol·h/L
Arm/Group | Test Cocktail (T) | Digoxin (R1)
Number analyzed (Participants) | 27 | 28
nmol·h/L | 17.668 (1.039) | 18.303 (1.039)
Statistical Analysis 1: Comparison: Test Cocktail (T) vs Digoxin (R1); This statistical analysis assess the effect of the other cocktail compounds in treatment T on the secondary outcome measure of treatment R1; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric mean ratio (T/R1) (%) = 96.53, 90% CI 2-sided [92.08 to 101.20], Standard Deviation 10.1 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Area Under the Curve of Furosemide From 0 Extrapolated to Infinity (AUC 0-∞)
Description: Area under the concentration-time curve of furosemide in plasma over the time interval from 0 extrapolated to infinity (AUC 0-∞). Standard error presented is actually geometric standard error.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol·h/L
Arm/Group | Test Cocktail (T) | Furosemide (R2)
Number analyzed (Participants) | 20 | 20
nmol·h/L | 156.382 (1.049) | 160.551 (1.052)
Statistical Analysis 1: Comparison: Test Cocktail (T) vs Furosemide (R2); This statistical analysis assess the effect of the other cocktail compounds in treatment T on the secondary outcome measure of treatment R2; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric mean ratio (T/R2) (%) = 97.40, 90% CI 2-sided [90.87 to 104.41], Standard Deviation 9.6 — [estimate comment as in outcome 3, analysis 1]

11. Secondary Outcome: Area Under the Curve of Metformin From 0 Extrapolated to Infinity (AUC 0-∞)
Description: Area under the concentration-time curve of metformin in plasma over the time interval from 0 extrapolated to infinity (AUC 0-∞). Standard error presented is actually geometric standard error.
Time Frame: as for outcome 5
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol·h/L
Arm/Group | Test Cocktail (T) | Metformin Hydrochloride (R3)
Number analyzed (Participants) | 28 | 29
nmol·h/L | 1290.928 (1.033) | 1324.078 (1.033)
Statistical Analysis 1: Comparison: Test Cocktail (T) vs Metformin Hydrochloride (R3); This statistical analysis assess the effect of the other cocktail compounds in treatment T on the secondary outcome measure of treatment R3; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric mean ratio (T/R3) (%) = 97.50, 90% CI 2-sided [93.58 to 101.58], Standard Deviation 8.9 — [estimate comment as in outcome 5, analysis 1]

12. Secondary Outcome: Area Under the Curve of Rosuvastatin From 0 Extrapolated to Infinity (AUC 0-∞)
Description: Area under the concentration-time curve of rosuvastatin in plasma over the time interval from 0 extrapolated to infinity (AUC 0-∞). Standard error presented is actually geometric standard error.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol·h/L
Arm/Group | Test Cocktail (T) | Rosuvastatin (R4)
Number analyzed (Participants) | 22 | 25
nmol·h/L | 97.385 (1.072) | 90.479 (1.069)
Statistical Analysis 1: Comparison: Test Cocktail (T) vs Rosuvastatin (R4); This statistical analysis assess the effect of the other cocktail compounds in treatment T on the secondary outcome measure of treatment R4; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric mean ratio (T/R4) (%) = 107.63, 90% CI 2-sided [97.04 to 119.39], Standard Deviation 19.4 — [estimate comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) occurring up to 192 hours after intake of trial drug administration in each treatment period were assigned to treatment.
Description: The treated set (TS) included all randomized subjects who were documented to have taken at least 1 dose of study drug.
Arm/Group | Digoxin (R1) | Furosemide (R2) | Metformin Hydrochloride (R3) | Rosuvastatin (R4) | Test Cocktail (T)
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/30 | 0/29 | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/30 | 1/29 | 1/29 | 3/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Digoxin (R1) (N=28) | Furosemide (R2) (N=30) | Metformin Hydrochloride (R3) (N=29) | Rosuvastatin (R4) (N=29) | Test Cocktail (T) (N=28)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Digoxin (R1) (N=28) | Furosemide (R2) (N=30) | Metformin Hydrochloride (R3) (N=29) | Rosuvastatin (R4) (N=29) | Test Cocktail (T) (N=28)
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes